CLINICAL TRIAL: NCT06573242
Title: Home-based Cardiac Rehabilitation for People Living With Heart Failure and Their Caregivers- The DK: REACH-HF Pilot Study
Brief Title: Home-based Cardiac Rehabilitation for People Living With Heart Failure and Their Caregivers- The DK:REACH-HF Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Signe Stelling Risom, Senior researcher, Herlev and Gentofte Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H-24031772
Record Dates: First submitted 2024-08-26; First posted 2024-08-27 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure
Keywords: rehabilitation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DK:REACH-HF (Experimental): 12 weeks of homebased cardiac rehabilitation for patients with heart failure and their caregivers
  Interventions: Other: Home-based cardiac rehabilitation for people living with Heart Failure and their caregivers

INTERVENTIONS:
Other: Home-based cardiac rehabilitation for people living with Heart Failure and their caregivers — Intervention DK:REACH-HF is a home-based 12-week CR program for people living with HF and their caregivers.

SUMMARY:
Background: Participation in cardiac rehabilitation (CR) is a strong recommendation of clinical guidelines for the management of heart failure (HF) because it is demonstrated to be a clinically effective and cost-effective intervention. Despite this, Danish data shows the uptake of CR is suboptimal (51%). A major barrier is that the traditional mode of CR provision is centre based. Travelling (time and cost), dislike of group exercise, and inconvenient timings are some key problems to participation. A potential solution is use of home-based programmes as an alternative to traditional CR.

A novel home-based programme for patients with HF and their caregivers (REACH-HF), developed in the United Kingdom has achieved improvements in quality of life and proven to be cost effective. The REACH-HF program is translated and adapted into a Danish context (DK: REACH-HF) and is now ready to be tested in a Danish setting.

The aim of this project is to improve the access and uptake of CR among HF patients in Denmark, particularly in subgroups of patients who currently do not benefit from center-based CR.

DETAILED DESCRIPTION:
Globally, Heart Failure (HF) is a common and severe disease affecting millions of people and a major driver of poor health-related quality of life (HRQoL), increased risk of hospitalization and high healthcare costs. Due to the aging of the population as well as the improvements of life-prolonging cardiovascular invasive and medical treatments, the prevalence of patients living with HF is increasing and as many as 1 in 5 people are expected to develop HF during their lifetime. Cardiac rehabilitation (CR) for people living with HF has been demonstrated to be clinically efficacious and cost-effective by improving HRQoL and reducing the risk of hospital readmission. Guidelines therefore strongly recommend CR for people living with HF. However, the uptake and provision of CR for people with HF in Denmark is suboptimal with only 51 % of HF patients participating. Furthermore, there is evidence of social inequality in both referral and participation rates. Reasons for low uptake are complex, but a major barrier is that traditional mode of CR provision is center based. Barriers to center-based programs for patients include travel time and costs and dislike of group sessions. A key potential solution is therefore greater use of alternative modes of CR delivery.

Developed in the UK, 'Rehabilitation EnAblement in CHronic Heart Failure' REACH-HF is an evidence- and theory-based, patient-centred self-care home-based support program co-developed with patients, caregivers, and clinicians to meet the above challenges. Evaluated in the multicenter randomized controlled trial, participation in the REACH-HF programme has shown improved HRQoL for patients with HF and to be cost-effective in a UK healthcare setting. Furthermore, caregivers increased their confidence in the caregiver role. The REACH-HF is now being rolled out routinely across the UK National Health Service, improving CR access for people with HF and their caregivers. Including the core components of comprehensive CR, the REACH-HF program aligns with Danish guidelines. As part of the DK:REACH-HF project, the REACH-HF program and its materials have been translated and adapted into a Danish context. This adaptation process included the consideration of contextual differences between the healthcare systems, legislation, and culture of UK and Denmark and was informed by interviews with leaders and experts in cardiology, healthcare professionals working with HF in both hospital and municipality settings, as well as caregivers and patients. Following this evidence-based approach, the DK:REACH-HF is now ready to be assessed for its feasibility and acceptability to inform wider implementation for Danish patients with HF and their caregivers.

To investigate the feasibility of the DK:REACH-HF program the investigators will employ a single-arm, pre-post mixed methods design with a parallel process evaluation across two-three sites in Denmark. This will involve hospital centers and where applicable local municipalities where the DK:REACH-HF program will be delivered as an alternative to usual care.

The investigators intend to recruit a total of 75 HF patients and their caregivers where applicable, who will each receive the DK:REACH-HF programme delivered by a team of one or two trained intervention-facilitators.

DK:REACH-HF is a home-based 12-week CR program for people living with HF and their caregivers.

Intervention: Patients (and where applicable, caregivers) will be provided with the DK: REACH-HF manuals or/and a digital mobile phone application (Mobile app: "Mit Liv" My Life, translated) based on their preference and consist of four core elements.

The "REACH-HF manual" for patients that includes a detailed information on how to live with HF including topics as: the understanding of what HF is, managing symptom monitoring, information about managing medications, managing breathlessness and anxiety, and a choice of two structured progressive exercise programmes (a walking or/and a chair-based programme).

A Patient "Progress Tracker": an interactive booklet designed to facilitate learning from experience to record daily physical activity, symptoms, weight, and fluid monitoring etc.

The" Family and Friends Resource": a manual for caregivers aimed to increase their understanding of HF and focus on their own physical and mental health and wellbeing.

A two-day course for facilitators who will tailor the intervention for patients and caregivers.

Quantitative data.

Given the pilot nature of the study, the focus of statistical analysis and data presentation will take a descriptive approach for baseline demographic and outcome data. Continuous data will be reported as means ± standard deviation or percentage. Categorical data will be reported as frequencies and percentages. Pre-post-differences in outcomes will be reported as means and 95% confidence intervals.

Qualitative data.

A semi structured interview guide will be used in the process evaluation and will focus on topics such as practical issues managing the DK:REACH-HF intervention program from both a facilitator and participant perspective, delivery of the intervention, participant experience of the intervention etc. The transcribed qualitative data will be coded using NVivo and analyzed using qualitative thematic analysis as described by Braun and Clark.

Mixed methods

The investigators will use both qualitative and quantitative data to gain a more complete and deeper understanding of issues relating to homebased CR for people living with HF and their caregivers as well as for health care providers included as facilitators in the study. By using a mixed methods approach to answer the aim of this research the investigators believe it can be examined in a more nuanced way.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years
* Confirmed diagnosis of Heart Failure (HF) with reduced Ejection Fraction (HFrEF) (Ejection Fraction (EF) <45%)
* No worsening of HF symptoms within past 2 weeks resulting in hospitalization (to ensure stable patients)
* Are deemed suitable for participating in Cardiac Rehabilitation (CR) by the outpatient HF clinic

Exclusion Criteria:

* Have undertaken CR within the past 12 months
* Are unwilling/unable to travel to a rehabilitation center in the municipality or at the hospital
* Are unable to understand the study information and/or corporate on giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Minnesota Living with Heart Failure questionnaire | 12 weeks
  Questionnaire. The MLHFQ is a disease-specific questionnaire for patients with Heart failure, comprising 21 items rated on six-point Likert scales, represening, from 0 (none) to 5 (very much). It provides a total score (range 0-105) Higher scores means worse health related quality of life (HRQoL).

SECONDARY OUTCOMES:
EQ-5D-5L | 12 weeks
  Generic Health related quality of life. Questionnaire. comprises five dimensions, describing different aspect of health: mobility, self-care, usual activities, pain / discomfort and anxiety / depression. Each dimension has five response levels: (1) no problems,(2) slight problems, (3) moderate problems, (4) severe problems, (5) unable to/extreme. Higher scores means worse generic health related quality of life.
Hospital Anxiety and Depression Scale (HADS) | 12 weeks
  Questionnaire. Minimum Value: 0 Maximum Value: 21 (for each subscale: anxiety and depression; the total score can range from 0 to 42) Higher Scores Mean: Worse anxiety or depression. HADS assesses levels of anxiety and depression through separate subscales for each condition
The European Heart Failure Self-care Behaviour Scale (EHFScB) | 12 weeks
  Questionnaire: comprising 12 items rated on a 5-point scale between 1 (I completely agree) and 5 (I completely disagree). Higher score means worse heart failure self-care behaviour
Kansas City cardiomyopathy questionnaire (KCCQ) | 12 weeks
  Questionnaire. The KCCQ-12 is a 12-item questionnaire that measures physical function, symptoms, social function, and quality of life. Each Item responses are coded in sequential order (1, 2, 3, etc.) from the worst to the best status. Higher score means better status.
Caregiver contribution to HF self-management | 12 weeks
  Questionnaire. The caregiver contribution to self-care consist of 10 items devided into 3 scales and uses a 4-point Likert scale (neveror rarely, sometimes, frequently, always or daily). Higher scores means higher contribution to self-care
Caregiver burden scale | 12 weeks
  Questionnaire. The Caregiver burden scale consist of 22 items devided into 5 scales and uses a 4 -point Likert scale rating from 1: "not at all" to 4: "very much". Higher scores means higher degree of burden.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Herlev and Gentofte HUniversity Hospital, Herlev, copenhagen
  - Herlev and Gentofte University Hospital, Herlev, Herlev

IPD SHARING:
Plan to Share IPD: Yes